CLINICAL TRIAL: NCT05548790
Title: Should Preoperative Information Before Impacted Third Molar Extraction Be Visual, Verbal or Both?
Brief Title: Should Preoperative Information Before Impacted Third Molar Extraction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Kevser SANCAK, oral and maxillofacial surgery, principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-2022-14
Record Dates: First submitted 2022-09-09; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Impacted Third Molar Tooth; Dental Anxiety
Keywords: third molar extraction; Dental anxiety; preoperative information

STUDY DESIGN:
Intervention Model Description: Group 1 was informed via silent video with subtitle, group 2 was informed via video with background audio, group 3 was informed with written information brochure, group 4 (control group) was informed verbally.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1: patients were given information via silent video with subtitle (5-minute)
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S); Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)
- Group 2 (Experimental): Group 2: patients were given information via video with background audio (5-minute 34-second)
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S); Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)
- Group 3 (Experimental): Group 3: patients were given written information brochure
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S); Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)
- Group 4 (Experimental): Group 4: patients were given information verbally
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S); Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)

INTERVENTIONS:
Behavioral: Spielberger State Anxiety Inventory (STAI-S) — STAI is one of the most frequently used scales in anxiety research, although it is not a specific scale for dental anxiety
Behavioral: Dental Fear Scale (DFS) — DFS is a scale developed by Kleinknecht used to determine dental fear in different dimensions. This is a Likert-type scale with a score of 1-5. It has 20 items. It examines the level of fear in terms of dentist avoidance, somatic symptoms of fear, and fear of various applications in dentistry practice
Behavioral: Modified Dental Anxiety Scale (MDAS) — MDAS was developed by Humphris et al. by adding a question related to injection. The scale consists of five-point Likert-type rating with five options. The scoring in this scale varies between 5 and 25
Behavioral: Visual Analog Scale (VAS) — VAS is ideal for evaluating situations that cannot be measured using digital and oral information. In the present study, a scale comprising 100-mm closed-end line was used to measure the anxiety level. One end of the scale was labeled as "no anxiety" and the other end as "maximum anxiety imaginable

SUMMARY:
The main objective of the present study was to evaluate the effects of different preoperative information techniques (verbal, written, video with background audio, and silent video with subtitles) on patients' anxiety levels before and after third molar extraction. The secondary objective was to determine the superiority of the information methods evaluated over each other. We hypothesized that the information provided by video with or without background audio would decrease preoperative and postoperative anxiety levels more effectively than information provided by verbal and written methods.

DETAILED DESCRIPTION:
This prospective study included 86 patients who underwent third molar extraction under local anesthesia in the Oral and Maxillofacial Department, Faculty of Dentistry, Ankara Yıldırım Beyazıt University, Turkey, between May and June 2022. The research protocol was approved by The Yıldırım Beyazıt University Oral and Health Training and Research Hospital Ethical Committee,Turkey. (No: E-2022-14) Spielberger State Anxiety Inventory (STAI-S), Dental Fear Scale (DFS), Modified Dental Anxiety Scale (MDAS), and Visual Analog Scale (VAS) are commonly used questionnaires for dental anxiety. The latter asked only about age and sex. They were used together before and immediately after surgery to obtain better results in this study.

After examining the panoramic radiographs, patients who underwent extraction were included in Classes 1 and II, Positions A and B according to Pell-Gregory classification, and mesioangular and vertical positions according to the Winter classification.

Each patient was examined by the researcher. The patients were informed about the procedure, and written informed consent was obtained from the patient's preoperative assessment clinic. If a patient had additional questions, they were included as part of the investigation Patients were assigned to 4 groups: Group 1 was informed via silent video with subtitle, group 2 was informed via video with background audio, group 3 was informed with written information brochure, group 4 (control group) was informed preoperatively verbally. The Spielberger State Anxiety Inventory (STAI-S), Dental Fear Scale (DFS), Modified Dental Anxiety Scale (MDAS), and visual analog scale (VAS) were used pre- and postoperatively to evaluate the dental anxiety of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not have pain
* Signs of infection related to the third molar were included
* American Society of Anesthesiologists physical status score I and II
* The absence of any systemic disease and regular medication use

Exclusion Criteria:

* Patients have the presence of an existing psychiatric disorder, psychiatric disorders, anxiolytic or antidepressant drug treatment
* Patients who were pregnant or lactated
* Patients who couldn't understand or fill out questionnaires, had presence of visual or auditory deficits, refuse to watch the video or join the study, had incomplete data
* Patients who had a previous negative experience with dental treatment were excluded from the study, as it may cause higher anxiety levels
* Those who watched a video on the subject before were not included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of anxiety with Spielberger State Anxiety Inventory(STAI-S) between groups preoperatively and postoperatively | 2 minutes
  STAI-S is a 20-item scale that determines the current anxiety level of the patient with reliability and validity in Turkish. Widely used to assess anxiety, the STAI explores the transient state of anxiety, and patients report how they are feeling at the current time point. It is scored using a 4-level frequency scale ranging from 0 to 3. The total score ranges from 20 to 80, higher scores indicates higher anxiety
Evaluation of anxiety with Dental Fear Survey(DFS) between groups preoperatively and postoperatively | 2 minutes
  DFS is which consists of 20-items is used to determine physiological responses to dental stimuli via a Likert-type scale ranging from 1 to 5. Total scores change from 20 to 100 point. It collects the evaluation of dental anxiety under 3 headings. The first 2 questions assess avoidance of dentistry, questions 3-7 show physiological arousal, and questions 8-20 predict fear of certain situations
Evaluation of anxiety with Modified Dental Anxiety Scale(MDAS) between groups preoperatively and postoperatively | 1 minute
  MDAS which is created by adding one question to the Corah Dental Anxiety Scale have 5-item questionnaire with 5-point Likert-type scale. Scale shows points between 5 and 25
Evaluation of anxiety with Visual Analog Scale (VAS) between groups preoperatively and postoperatively | 1 minute
  VAS is a digital and verbal assessment scale used to measure anxiety. A closed-ended scale of 0-100 mm ("0" no anxiety, "100" maximum imaginable anxiety) was used in the study, and participants were asked to put a mark on the VAS scale, which they thought showed the degree of their current anxiety

CONTACTS AND LOCATIONS:
Overall Officials: kevser sancak, Principal Investigator — Ankara Yıldırım Beyazıt University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım beyazıt University, Faculty of Dentistry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Muglali M, Komerik N. Factors related to patients' anxiety before and after oral surgery. J Oral Maxillofac Surg. 2008 May;66(5):870-7. doi: 10.1016/j.joms.2007.06.662. PMID 18423273
- [Background] Laskin DM, Priest JH, Alfaqih S, Carrico CK. Does Viewing a Third Molar Informed Consent Video Decrease Patients' Anxiety? J Oral Maxillofac Surg. 2018 Dec;76(12):2515-2517. doi: 10.1016/j.joms.2018.08.001. Epub 2018 Aug 15. PMID 30193118
- [Background] Sirin Y, Humphris G, Sencan S, Firat D. What is the most fearful intervention in ambulatory oral surgery? Analysis of an outpatient clinic. Int J Oral Maxillofac Surg. 2012 Oct;41(10):1284-90. doi: 10.1016/j.ijom.2012.06.013. Epub 2012 Jul 23. PMID 22832662
- [Background] de Jongh A, Olff M, van Hoolwerff H, Aartman IH, Broekman B, Lindauer R, Boer F. Anxiety and post-traumatic stress symptoms following wisdom tooth removal. Behav Res Ther. 2008 Dec;46(12):1305-10. doi: 10.1016/j.brat.2008.09.004. Epub 2008 Sep 25. PMID 18954863